CLINICAL TRIAL: NCT01320215
Title: Complications Associated With Promontofixation for Pelvic Organ Prolapse: a Randomized Trial Comparing Robot Assisted Laparoscopic and Non-robot Assisted Laparoscopic Surgical Procedures
Brief Title: Complications Associated With Promontofixation for Pelvic Organ Prolapse: Comparing Robot Assisted Laparoscopic and Non-robot Assisted Laparoscopic Surgical Procedures
Acronym: RoboLaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRC-N/2010/SD-01; 2010-A01110-39 (Other: ANSM)
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: da Vinci Robot; uterine prolapse; vaginal prolapse; sacrohysteropexy
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot arm (Experimental): The patients in this arm will have a robot-assisted promontofixation.
  Interventions: Procedure: Robot-assisted promontofixation
- Non-robot arm (Active Comparator): The patients in this arm with have a promotofixation via a laparoscopy, but without robot assistance.
  Interventions: Procedure: Non-robot assisted promontofixation

INTERVENTIONS:
Procedure: Robot-assisted promontofixation — Sacrohysteropexy with robotic assistance (da Vinci robot)
  Arms: Robot arm
Procedure: Non-robot assisted promontofixation — Laparoscopic sacrohysteropexy, without robot assistance
  Arms: Non-robot arm

SUMMARY:
The primary objective of this study is to compare 30-day complication rates associated with promontofixation for pelvic organ prolapse performed via a robot-assisted laparoscopic technique versus a non-robot-assisted laparoscopic technique. Secondary objectives include comparing technical data, anatomical correction, prolapse recurrence, incontinence, quality of life and medico-economic data between the two techniques.

The patient diary did not allow the collection of sufficiently precise data to meet the secondary medico-economic objective of the study. Access to data from the National Health Data System (SDNS), which was not available at the time of the initial drafting of this protocol, now makes it possible to obtain a complete picture of patients' health care consumption. We propose, therefore, to extract data from the SNIIRAM via the SNDS (matching of patients' NIR to their health care consumption) in order to retrieve and accurately estimate the cost of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a first,(primo-event), symptomatic, genito-urinary prolapse of at least stage II (POP-Q classification) requiring surgery
* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 60 months of follow-up

Exclusion Criteria:

* The patient is participating in another study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* Patient has a stage-1 prolapse (POP-Q classification)
* Patient has asymptomatic prolapse
* The patient has a prolapse recurrence (i.e. this is not the first case of prolapse)
* The patient is not available for 60 months of follow-up
* Patient has a vaginal or urinary infection
* Patient has poorly-adjusted diabetes
* Patient on long-term corticotherapy
* Patient has previously had pelvic radiotherapy
* Patient has contraindication for anesthesia
* Patient has an intestinal inflammatory disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2011-06-22 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
presence/absence of complications (composite score) | 30 days
  The occurrence (in the per-operative phase or within 30 days post-op) of at least one of the following: 1) bleeding complications: hemoperitoneum, blood loss> = 500 ml, transfusion; 2) infectious complications: wound infection, abscess, discitis, mesh infection; 3) any wound caused by a surgeon movement: bladder, digestive, ureteral, or vascular injuries; (4) medical complications: deep vein thrombosis, pulmonary embolism, pneumopathy; 5) trocart sites: infection, hernia; 6) conversion to a laparoscopic or open surgical technique not related to pre-existing adhesions; 7) reintervention; 8) neurological complications: neurological disorders, complications of the central neurological system, sciatica; 9) others: complete urinary retention, lower urinary tract infection, extrusion, erosion of the mesh, hospitalization in intensive care; 10) death.

SECONDARY OUTCOMES:
Time needed to prep the operation room (min) | 1 day
length of hospital stay (days) | 1 month
  The number of days the patient stays in the hospital following promontofixation
Operative time (min) | 1 day
  The time elapsed between incision and closure of the patient
Anesthesia time (min) | 1 day
  The time elapsed between anethesia induction and awakening
Equipment installation time (min) | 1 day
  Time elapsed between installation of trocarts and insertion of endoscopic instruments (robot arms or coelioscopic tools)
Surgical time (min) | 1 day
  The time spent manipulating endoscopic intruments or console time for robotic techniques.
Presence/absence of conversion | Day 1
  In the robot arm: the need to convert to laparoscopic procedure or open procedure; in the non-robot arm: the need to convert to an open procedure
presence/absence of a re-intervention | 30 days
Presence/absence of urinary incontinence | 3 months
Presence/absence of urinary incontinence | 12 months
Presence/absence of urinary incontinence | 36 months
Presence/absence of urinary incontinence | 60 months
presence/absence of constipation | 3 months
presence/absence of constipation | 12 months
presence/absence of constipation | 36 months
presence/absence of constipation | 60 months
Presence/absence of fecal incontinence | 3 months
Presence/absence of fecal incontinence | 12 months
Presence/absence of fecal incontinence | 36 months
Presence/absence of fecal incontinence | 60 months
presence/absence of dysparunia | 3 months
presence/absence of dysparunia | 12 months
presence/absence of dysparunia | 36 months
presence/absence of dysparunia | 60 months
POP-Q score | 3 months
POP-Q score | 12 months
POP-Q score | 36 months
POP-Q score | 60 months
Urodynamic exam Q max (ml/s) | 3 months
  Urination rate il ml/s
Urodynamic exam Q max (ml/s) | 12 months
  Urination rate il ml/s
Urodynamic exam Q max (ml/s) | 36 months
  Urination rate il ml/s
Urodynamic exam Q max (ml/s) | 60 months
  Urination rate il ml/s
Urodynamic exam, volume urinated (ml) | 3 months
  the volume urinated in ml
Urodynamic exam, volume urinated (ml) | 12 months
  the volume urinated in ml
Urodynamic exam, volume urinated (ml) | 36 months
  the volume urinated in ml
Urodynamic exam, volume urinated (ml) | 60 months
  the volume urinated in ml
Urodynamic exam: post-mictionnel residu (ml) | 3 months
Urodynamic exam: post-mictionnel residu (ml) | 12 months
Urodynamic exam: post-mictionnel residu (ml) | 36 months
Urodynamic exam: post-mictionnel residu (ml) | 60 months
Urodynamic exam: fonctional bladder capacity (ml) | 3 months
  bladder capacity in ml
Urodynamic exam: fonctional bladder capacity (ml) | 12 months
  bladder capacity in ml
Urodynamic exam: fonctional bladder capacity (ml) | 36 months
  bladder capacity in ml
Urodynamic exam: fonctional bladder capacity (ml) | 60 months
  bladder capacity in ml
Urodynamic exam: urethral closure pressure (cm water) | 3 months
  urethral closure pressure in cm of water
Urodynamic exam: urethral closure pressure (cm water) | 12 months
  urethral closure pressure in cm of water
Urodynamic exam: urethral closure pressure (cm water) | 36 months
  urethral closure pressure in cm of water
Urodynamic exam: urethral closure pressure (cm water) | 60 months
  urethral closure pressure in cm of water
Wexner anal incontinence score | 3 months
Wexner anal incontinence score | 12 months
Wexner anal incontinence score | 36 months
Wexner anal incontinence score | 60 months
ODS constipation score | 3 months
ODS constipation score | 12 months
ODS constipation score | 36 months
ODS constipation score | 60 months
Visual analog scale for pain | day 1
Visual analog scale for pain | day 2
Visual analog scale for pain | day 3
Visual analog scale for pain | day 4
Visual analog scale for pain | 3 months
Visual analog scale for pain | 12 months
Visual analog scale for pain | 36 months
Visual analog scale for pain | 60 months
Patient satisfaction | Day 4
  Is the patient very satisfied, satisfied, somewhat unsatisfied, or very unsatisfied in relation to the procedure?
Patient satisfaction | 3 months
  Is the patient very satisfied, satisfied, somewhat unsatisfied, or very unsatisfied in relation to the procedure?
Patient satisfaction | 12 months
  Is the patient very satisfied, satisfied, somewhat unsatisfied, or very unsatisfied in relation to the procedure?
Patient satisfaction | 36 months
  Is the patient very satisfied, satisfied, somewhat unsatisfied, or very unsatisfied in relation to the procedure?
Patient satisfaction | 60 months
  Is the patient very satisfied, satisfied, somewhat unsatisfied, or very unsatisfied in relation to the procedure?
Questionnaire PFDI-20 | 3 months
Questionnaire PFDI-20 | 12 months
Questionnaire PFDI-20 | 36 months
Questionnaire PFDI-20 | 60 months
Questionnaire PFIQ-7 | 3 months
Questionnaire PFIQ-7 | 12 months
Questionnaire PFIQ-7 | 36 months
Questionnaire PFIQ-7 | 60 months
Questionnaire PISQ-12 | 3 months
Questionnaire PISQ-12 | 12 months
Questionnaire PISQ-12 | 36 months
Questionnaire PISQ-12 | 60 months
Questionnaire SF36 | 3 months
Questionnaire SF36 | 12 months
Questionnaire SF36 | 36 months
Questionnaire SF36 | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Droupy, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (18):
- France (18):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - Groupe Urologie Saint Augustin, Bordeaux
  - APHP - Centre Hospitalier Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nancy - Hôpitaux de Brabois, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice - Hôpitaux L'Archet 1 et 2, Nice
  - Clinique Kennedy, Nîmes
  - Groupe Hospitalier Diaconesses Croix Saint-Simon - Site Reuilly, Paris
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - CHU de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital PontChaillou, Rennes
  - Clinique Belledonne, Saint Martin d'Héres
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg
  - Hôpital Foch, Suresnes
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse
  - CHRU de Tours - Hôpital Bretonneau, Tours

REFERENCES:
- [Result] Gris JC, Chea M, Bouvier S, Pereira FR. Antiphospholipid Antibodies in Mental Disorders. Semin Thromb Hemost. 2025 Jun;51(4):448-456. doi: 10.1055/s-0044-1788696. Epub 2024 Jul 24. PMID 39047993